CLINICAL TRIAL: NCT07384494
Title: High-Flow Nasal Cannula Versus Conventional Oxygen to Prevent Hypoxaemia During Awake Tracheal Intubation: A Multicentre, Open-Label, Randomised Controlled Trial (OXYOPTI-ATI)
Brief Title: High-flow Nasal Cannula Versus Conventional Oxygen During Awake Tracheal Intubation With Difficult Airways
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wenxian Li (Other)
Responsible Party: Sponsor-Investigator, Wenxian Li, Professor and Chief Physician, Department of Anesthesiology, Eye & ENT Hospital of Fudan University, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EENTFudan 2025155-1
Record Dates: First submitted 2026-01-20; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Awake Tracheal Intubation; Difficult Airway
Keywords: Awake tracheal intubation; High-flow nasal cannula; Difficult airway; hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HFNC group (Experimental): During awake tracheal intubation, participants receive heated and humidified high-flow nasal cannula oxygen therapy at a flow rate of 40 L/min, FiO₂ of 100%, and a temperature of 37 °C, starting before the procedure and continuing until successful intubation is confirmed by the presence of end-tidal carbon dioxide.
  Interventions: Device: High-Flow Nasal Cannula
- LFNC group (Active Comparator): During awake tracheal intubation, participants receive oxygen via a disposable nasal cannula at a flow rate of 4 L/min, starting before the procedure and continuing until successful intubation is confirmed by the presence of end-tidal carbon dioxide.
  Interventions: Device: Ligh-Flow Nasal Cannula

INTERVENTIONS:
Device: High-Flow Nasal Cannula — A heated and humidified high-flow nasal oxygen therapy device（Fisher & Paykel，East Tamaki，New Zealand） set at a flow rate of 40 L/min, an inspired oxygen fraction (FiO₂) of 100%, and a temperature of 37 °C.
  Arms: HFNC group
Device: Ligh-Flow Nasal Cannula — Low-flow oxygen delivered via a disposable nasal cannula at a flow rate of 4 L/min.
  Arms: LFNC group

SUMMARY:
Study Background Airway management is one of the most fundamental and critical technical procedures in anesthesiology, critical care, and emergency medicine. Difficult airway management remains a major challenge in these fields, particularly when a "cannot intubate, cannot ventilate" scenario occurs during the induction of general anesthesia. Such events can rapidly lead to hypoxemia, resulting in brain injury or even death, and have become a significant source of anesthesia-related severe complications and medical disputes.

Awake tracheal intubation (ATI) is considered the gold standard for airway management in patients with anticipated difficult airways, as it preserves spontaneous breathing and thereby reduces the risk of catastrophic airway failure during anesthesia induction. However, despite routine supplemental oxygen administration, hypoxemia remains one of the most common and potentially serious complications during ATI. When low-flow oxygen therapy (<30 L/min) is used, the reported incidence of hypoxemia (SpO₂ ≤ 90%) ranges from 12% to 29%. Once hypoxemia occurs during ATI, it may not only interrupt the procedure, increase the number of intubation attempts, and reduce the likelihood of successful intubation, but also trigger serious cardiovascular events, thereby compromising patient safety.

High-flow nasal cannula (HFNC) oxygen therapy can deliver heated and humidified gas at flow rates of up to 70 L/min and improve oxygenation and ventilation through mechanisms such as anatomical dead space washout, reduction of work of breathing, and generation of continuous positive airway pressure. HFNC has been shown to improve oxygenation in a variety of medical and procedural settings. However, evidence regarding the role of HFNC during awake tracheal intubation remains controversial and of low quality. There is an urgent need for well-designed multicenter randomized controlled trials specifically focused on the ATI setting, using hypoxemic events as the primary outcome and applying strictly standardized procedures, to provide high-quality evidence on the effectiveness and safety of HFNC during ATI. Such evidence is essential to inform clinical practice and support future updates of airway management guidelines.

Study Hypothesis This study hypothesizes that, in patients with anticipated difficult airways undergoing ATI, HFNC is more effective in preventing intubation-related hypoxemic events than conventional low-flow nasal cannula oxygen therapy.

Study Objectives

Primary Objective:

To evaluate the effectiveness of high-flow nasal cannula oxygen therapy compared with conventional low-flow nasal cannula oxygen therapy in preventing hypoxemia during ATI in patients with anticipated difficult airways.

Secondary Objectives:

To assess the effects of high-flow nasal cannula oxygen therapy versus conventional low-flow nasal cannula oxygen therapy on procedural outcomes of awake tracheal intubation, including the rate of interventions required after hypoxemia, first-attempt intubation success rate, number of intubation attempts, overall ATI success rate, intubation time, and the incidence of adverse events.

Study Methods This study is a multicenter, randomized controlled clinical trial. Adult patients undergoing ATI will be recruited from six tertiary hospitals in China. Participants will be randomly assigned to receive either high-flow nasal cannula oxygen therapy or conventional low-flow nasal cannula oxygen therapy throughout the intubation procedure. The study will compare the incidence of hypoxemia between the two groups and further evaluate intubation success rates, intubation time, the need for rescue interventions following hypoxemia, and the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an anticipated difficult airway;
* Planned awake tracheal intubation;
* Age ≥ 18 years;
* Willingness to participate in the study and provision of written informed consent.

Exclusion Criteria:

* Contraindications to HFNC use, such as severe nasal obstruction or deformity, recent (within 3 months) nasal or skull base surgery, skull base fracture, or active epistaxis;
* Hemodynamic instability, defined as a mean arterial pressure (MAP) < 65 mmHg or the need for vasoactive medications to maintain blood pressure;
* Pregnancy;
* Current participation in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemia（SpO₂≤ 90%） | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.

SECONDARY OUTCOMES:
Incidence of SpO₂ ≤ 80% | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
Lowest SpO₂ | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
Cumulative duration of hypoxemia | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
Area under the curve (AUC) for SpO₂ ≤ 90% | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
Number of hypoxemic episodes per participant (defined as the first occurrence of SpO₂ ≤ 90% after preoxygenation counted as one episode; subsequent episodes counted if SpO₂ returns to normal and then decreases again) | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
SpO₂ at the time of successful intubation | At the time of successful intubation up to 24 hours
End-tidal carbon dioxide (EtCO₂) at the time of successful intubation | At the time of successful intubation up to 24 hours
Proportion of participants requiring rescue interventions after the occurrence of hypoxemia | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
First-attempt intubation success rate | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
Awake tracheal intubation success rate | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
Intubation time | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.
  Defined as the duration from initiation of ATI to confirmation of successful intubation by end-tidal carbon dioxide
Incidence of adverse events | From initiation of awake tracheal intubation to completion of successful tracheal intubation confirmed by end-tidal carbon dioxide (EtCO₂), assessed up to 30 minutes.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Wuwei People's Hospital, Wuwei, Gansu
  - South China Hospital of Shenzhen University, Shenzhen, Guangzhou
  - Baoding No.1 Central Hospital, Baoding, Hebei
  - Pizhou Hospital of Traditional Chinese Medicine, Pizhou, Jiangsu
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First People's Hospital of Neijiang, Neijiang, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cascio RS, Kilmon CA. Pervasive developmental disorder, not otherwise specified: primary care perspectives. Nurse Pract. 1997 Jul;22(7):11, 15-6, 18 passim. PMID 9253013
- [Background] Law JA, Morris IR, Brousseau PA, de la Ronde S, Milne AD. The incidence, success rate, and complications of awake tracheal intubation in 1,554 patients over 12 years: an historical cohort study. Can J Anaesth. 2015 Jul;62(7):736-44. doi: 10.1007/s12630-015-0387-y. Epub 2015 Apr 24. PMID 25907462
- [Background] Ho AM, Chung DC, To EW, Karmakar MK. Total airway obstruction during local anesthesia in a non-sedated patient with a compromised airway. Can J Anaesth. 2004 Oct;51(8):838-41. doi: 10.1007/BF03018461. PMID 15470176
- [Background] Badiger S, John M, Fearnley RA, Ahmad I. Optimizing oxygenation and intubation conditions during awake fibre-optic intubation using a high-flow nasal oxygen-delivery system. Br J Anaesth. 2015 Oct;115(4):629-32. doi: 10.1093/bja/aev262. Epub 2015 Aug 7. PMID 26253608
- [Background] Vourc'h M, Huard D, Le Penndu M, Deransy R, Surbled M, Malidin M, Mahe PJ, Guitton C, Roquilly A, Malard O, Feuillet F, Rozec B, Asehnoune K. High-flow oxygen therapy versus facemask preoxygenation in anticipated difficult airway management (PREOPTI-DAM): an open-label, single-centre, randomised controlled phase 3 trial. EClinicalMedicine. 2023 May 22;60:101998. doi: 10.1016/j.eclinm.2023.101998. eCollection 2023 Jun. PMID 37251624
- [Background] Mangan CE, Borow L, Burtnett-Rubin MM, Egan V, Giuntoli RL, Mikuta JJ. Pregnancy outcome in 98 women exposed to diethylstilbestrol in utero, their mothers, and unexposed siblings. Obstet Gynecol. 1982 Mar;59(3):315-9. PMID 7078877
- [Background] Kinsella SM, Winton AL, Mushambi MC, Ramaswamy K, Swales H, Quinn AC, Popat M. Failed tracheal intubation during obstetric general anaesthesia: a literature review. Int J Obstet Anesth. 2015 Nov;24(4):356-74. doi: 10.1016/j.ijoa.2015.06.008. Epub 2015 Jun 30. PMID 26303751
- [Background] Heidegger T. Management of the Difficult Airway. N Engl J Med. 2021 May 13;384(19):1836-1847. doi: 10.1056/NEJMra1916801. No abstract available. PMID 33979490
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488